CLINICAL TRIAL: NCT06980636
Title: Shengmai Liquid for Long COVID Fatigue: a Randomized Placebo-controlled Trial.
Brief Title: A Trial of Shengmai Liquid for Long COVID Fatigue.
Acronym: Shengmai LOFT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing University of Chinese Medicine (Other)
Collaborators: Institute of Chemistry - Vietnam Academy of Science and Technology (Unknown); Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Huijuan Cao, Professor, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023YFE0198400; 2023YFE0198400 (Other Grant/Funding Number: Ministry of Science and Technology of the People´s Republic of China)
Record Dates: First submitted 2025-05-18; First posted 2025-05-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-06

CONDITIONS: Long COVID Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shengmai Liquid (Experimental): For patients with Long COVID characterized by persistent fatigue who meet the inclusion and exclusion criteria, 100 patients will be randomly divided into a Shengmaiyin treatment group and a placebo control group using a random method. The Shengmaiyin treatment group will be given the traditional Chinese medicine Shengmaiyin oral liquid (produced by Jilin Aodong Yanbian Pharmaceutical Co., Ltd., with the approval number Z41021384. Ingredients: Codonopsis pilosula, Ophiopogon japonicus, Schisandra chinensis, excipients: sucrose, sodium benzoate, ethylparaben, specification 10m1/bottle), taken orally at a dose of 10ml per time, three times a day
  Interventions: Drug: Shengmai Liquid
- Placebo (Placebo Comparator): The placebo group will be given a simulated Shengmaiyin oral liquid (provided by Jilin Aodong Yanbian Pharmaceutical Co., Ltd., with main ingredients water, brown sugar, flavoring agents, etc., specification 10m/bottle), 10ml per time, three times a day. The treatment course for Shengmaiyin or placebo will be 8 weeks (56 days), with follow-up continuing until 30 days after the end of the treatment course.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Shengmai Liquid — The Shengmaiyin treatment group will be given the traditional Chinese medicine Shengmaiyin oral liquid (produced by Jilin Aodong Yanbian Pharmaceutical Co., Ltd., with the approval number Z41021384. Ingredients: Codonopsis pilosula, Ophiopogon japonicus, Schisandra chinensis, excipients: sucrose, sodium benzoate, ethylparaben, specification 10m1/bottle), taken orally at a dose of 10ml per time, three times a day
  Arms: Shengmai Liquid
Other: Placebo — A simulated Shengmaiyin oral liquid (provided by Jilin Aodong Yanbian Pharmaceutical Co., Ltd., with main ingredients water, brown sugar, flavoring agents, etc., specification 10m/bottle), 10ml per time, three times a day. The treatment course for Shengmaiyin or placebo will be 8 weeks (56 days), with follow-up continuing until 30 days after the end of the treatment course.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if Shengmai liquid works to treat Long Covid fatigue. It will also learn about the safety of Shengmai liquid. The main questions it aims to answer are:

* Dose the Shengmai liquid will reduce the level of fatigue in the participants and reduce the fatigue scale score of the participants?
* Dose the Shengmai liquid will reduce the level of anxiety and depression in the participants and improve the sleep quality and quality of life of the participants Researchers will compare Shengmai oral liquid to a placebo (a look-alike substance that contains no drug) to see if Shengmai liquid works to treat Long Covid fatigue.

Participants will:

* Take Shengmai liquid or a placebo every day for 8 weeks.
* Visit the clinic once every 4 weeks for check up and test. There are a total of two telephone follow-ups, one follow-up 15 days after the treatment starts and another follow-up 30 days after the treatment ends.
* Participants' medication responses and scale scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75 years;
* Meet the above diagnostic criteria;
* Meet the traditional Chinese medicine syndrome diagnostic criteria;
* Consent and sign the informed consent form

Exclusion Criteria:

* Currently in need of or expected to require high-flow oxygen therapy, positive pressure ventilation, invasive mechanical ventilation, or extracorporeal membrane oxygenation (ECMO) and other advanced respiratory support measures;
* Have a known history of active liver disease (excluding non-alcoholic fatty liver changes), including active hepatitis B or C infection, primary biliary cirrhosis, Child-Pugh class B or C liver function impairment, or acute liver failure. Liver function at screening shows any of the following: serum alanine aminotransferase (ALT) >3× the upper limit of normal (ULN); serum aspartate aminotransferase (AST) >3×ULN; serum bilirubin >2×ULN;
* Undergoing dialysis treatment, or known to have moderate to severe renal impairment (i.e., an estimated glomerular filtration rate (eGFR) value calculated based on serum creatinine using the CKD-EPI formula ≤45 mL/min/1.73 m² within 6 months before screening);
* Moderate to severe congestive heart failure within 6 months before screening (according to the New York Heart Association classification criteria, with cardiac function class III or IV), experienced a stroke, myocardial infarction, or coronary artery stent implantation; or have uncontrolled hypertension (defined as systolic blood pressure exceeding 160 mmHg or diastolic blood pressure exceeding 100 mmHg, with relevant records). Significant or clinically relevant electrocardiogram abnormalities, such as second-degree type II atrioventricular block, left bundle branch block, etc.;
* Suffered from influenza A, influenza B, or other infectious diseases within 3 months before screening;
* Have/ever had severe neurological diseases (epilepsy, convulsions, or seizures) or mental illness, or have a family history of mental illness;
* Pregnant or breastfeeding. Women who are breastfeeding or have a positive pregnancy test before taking the medication;
* History of malignant tumors within 5 years before screening, with existing and progressing tumors, and patients who are expected to need treatment during the study period;
* Have chronic fatigue syndrome or autoimmune diseases (such as rheumatoid arthritis, systemic lupus erythematosus, etc.);
* Known allergy to any component of the study drug;
* Diseases judged by the investigator to be unsuitable for participation in this study;
* Taken traditional Chinese medicine containing Codonopsis pilosula, Ophiopogon japonicus, Schisandra chinensis, or Astragalus membranaceus within 2 weeks before screening;
* Participating in other drug or medical device-related studies at the same time

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The degree of improvement in patient fatigue, measured using the Modified Fatigue Impact Scale (MFIS) | From enrollment to the end of follow up at 12 weeks
  MFIS is a standardized questionnaire reflecting physical and mental fatigue, consisting of 21 questions. Each question has five options (none at all, a little, sometimes, often, almost always), with a total score range of 0 to 84. The higher the score, the higher the degree of chronic fatigue.

SECONDARY OUTCOMES:
Traditional Chinese Medicine Syndrome Score Scale | From enrollment to the end of treatment at 8 week
  Measured once during the screening period before the start of the trial, and then at 30 days and 60 days during the trial, for a total of three measurements.
Improvement in depression, assessed using the 17-item Hamilton Depression Scale | From enrollment to the end of treatment at 8 weeks
  Measured once during the screening period before the start of the trial, and then at 30 days and 60 days during the trial, for a total of three measurements.
Improvement in anxiety, assessed using the Hamilton Anxiety Scale (HAMA) | From enrollment to the end of treatment at 8 weeks
  Measured once during the screening period before the start of the trial, and then at 30 days and 60 days during the trial, for a total of three measurements.
Improvement in sleep quality, assessed using the Pittsburgh Sleep Quality Index (PSQI) | From enrollment to the end of treatment at 8 week
  Measured once during the screening period before the start of the trial, and then at 30 days and 60 days during the trial, for a total of three measurements.
Improvement in quality of life, assessed using the World Health Organization Quality of Life Scale | From enrollment to the end of treatment at 8 weeks
  measured once during the screening period before the start of the trial, and then at 30 days and 60 days during the trial, for a total of three measurements.
six minute walk test（6MWT） | From enrollment to the end of treatment at 8 weeks
  Measured once during the screening period before the start of the trial, and then at 30 days and 60 days during the trial, for a total of three measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Di Tan Hospital, , Capital Medical University, Beijing, China, China

IPD SHARING:
Plan to Share IPD: Undecided